CLINICAL TRIAL: NCT01630278
Title: Impact of Early Targeted Ibuprofene Treatment of Patent Ductus Arteriosus (PDA) on Long Term Neurodevelopmental Outcome in Very Premature Infants (TRIOCAPI)
Brief Title: Early Ibuprofen Treatment of Patent Ductus Arteriosus (PDA) in Premature Infants (TRIOCAPI)
Acronym: TRIOCAPI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BRD/10/06-O
Record Dates: First submitted 2012-06-11; First posted 2012-06-28 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Patent Ductus Arteriosus
Keywords: Prematurity; patent ductus arteriosus; ibuprofen
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Small ductus (No Intervention)
- Large ductus ibuprofen (Experimental): Very premature infants with a large ductus, selected by an early echocardiogram, will receive ibuprofen before 12 hours of life
  Interventions: Drug: Ibuprofen
- Large ductus placebo (Placebo Comparator): Very premature infants with a large ductus, selected by an early echocardiogram, will receive placebo before 12 hours of life
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — Very premature infants with a large ductus, selected by an early echocardiogram, will receive ibuprofen before 12 hours of life
  Arms: Large ductus ibuprofen
Drug: Placebo — Very premature infants with a large ductus, selected by an early echocardiogram, will receive placebo before 12 hours of life
  Arms: Large ductus placebo

SUMMARY:
Very premature infants with a large ductus, selected by an early echocardiogram, will receive either ibuprofen or placebo before 12 hours of life. Follow-up will include repeated echocardiograms and cranial ultrasound at 36 hours, 14 days and 36 weeks of postconceptional age. The primary outcome will be survival without cerebral palsy at years.

ELIGIBILITY:
Inclusion Criteria:

* Gestational less than 28 weeks
* Postnatal age less than 12 hours

Max Age: 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 363 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
2-year survival without cerebral palsy | 2 years

SECONDARY OUTCOMES:
ASQ (Ages and Stages Questionnaire) score at 2 years | 2 years
Incidence of other prematurity-related morbidities (pulmonary, digestive, neurological, renal) | 2 years
  To compare the outcome between the large and the small ductus groups
Comparison of outcome according to the McNamara stage at surgical ligation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe ROZE, Professor, Study Chair — Nantes University Hospital
Locations (11):
- France (11):
  - University Hopsital, Angers
  - University Hopsital, Bordeaux
  - University Hospital, Créteil
  - University Hospital, Grenoble
  - University Hospital, Lille
  - University Hospital, Marseille
  - Univesity Hospital, Montpellier
  - University Hospital, Nantes
  - University Hospital (AP-HP Groupe hospitalier), Paris
  - University Hospital, Rennes
  - University Hospital, Tours

REFERENCES:
- [Derived] Roze JC, Cambonie G, Le Thuaut A, Debillon T, Ligi I, Gascoin G, Patkai J, Beuchee A, Favrais G, Flamant C, Durrmeyer X, Clyman R. Effect of Early Targeted Treatment of Ductus Arteriosus with Ibuprofen on Survival Without Cerebral Palsy at 2 Years in Infants with Extreme Prematurity: A Randomized Clinical Trial. J Pediatr. 2021 Jun;233:33-42.e2. doi: 10.1016/j.jpeds.2020.12.008. Epub 2020 Dec 9. PMID 33307111
- [Derived] Mitra S, Scrivens A, von Kursell AM, Disher T. Early treatment versus expectant management of hemodynamically significant patent ductus arteriosus for preterm infants. Cochrane Database Syst Rev. 2020 Dec 10;12(12):CD013278. doi: 10.1002/14651858.CD013278.pub2. PMID 33301630